CLINICAL TRIAL: NCT04679623
Title: Phase 1, Open-Label, Comparison Study to Evaluate the Safety and Pharmacokinetics of a Single Intramuscular Administration of 10 mg Midazolam Using an Auto-Injector vs Marketed Midazolam Vials in Healthy Adults.
Brief Title: Study of Midazolam in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rafa Laboratories (Industry)
Collaborators: Alachua Government Services, Inc. (Industry); Joint Project Management Office for Chemical, Biological, Radiological, and Nuclear Medical (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RLM-559-01
Record Dates: First submitted 2020-12-15; First posted 2020-12-22 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Status Epilepticus
MeSH Terms: conditions — Status Epilepticus | interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Midazolam Injection (Experimental): Midazolam injection, 10 mg
  Interventions: Combination Product: Midazolam
- Seizalam™ (Active Comparator): Seizalam, 10 mg
  Interventions: Drug: Seizalam

INTERVENTIONS:
Combination Product: Midazolam — Midazolam Injection, 10mg
  Arms: Midazolam Injection
Drug: Seizalam — Seizalam, 10 mg
  Arms: Seizalam™

SUMMARY:
This study is a phase 1, open-label, crossover, comparison study to evaluate the safety and pharmacokinetics (PK) of a single IM administration of 10 mg midazolam using Rafa's auto-injector compared with seizalam in healthy adults. All subjects will participate in both study periods which will span 28 days following a pre study screening visit.

ELIGIBILITY:
Inclusion Criteria:

1. Can understand and provide signed informed consent
2. Is a healthy male or healthy, non-pregnant, non-lactating female whose screening, physical exam, labs, vitals, and ECG are within normal range
3. Has a willingness to comply and be available for all protocol procedures
4. Is between age 18 and 55 years, inclusive on the day of injection
5. If the subject is female and of childbearing potential, she has a negative serum pregnancy test at screening and negative urine test within 24 hours prior to injection Note: A woman is considered of childbearing potential unless post-menopausal (≥ 1 year without menses) or surgically sterilized via bilateral oophorectomy, or hysterectomy or bilateral tubal ligation or successful Essure placement with documented confirmation test at least 3 months after the procedure
6. If the subject is female and of childbearing potential, she agrees to practice abstinence from sexual intercourse with men or use acceptable contraception up to 1 month after the end of study visit Note: Acceptable contraception methods are restricted to effective devices (approved oral contraceptives, Intrauterine Contraceptive Devices, NuvaRing®)
7. If the subject is male, he agrees to practice abstinence from sexual intercourse with women or use acceptable contraception up to 1 month after the end of study visit
8. Has a body mass index (BMI) ≥18.0 and ≤26.0 kg/m2 at screening
9. Has a negative urine drug screen
10. Has a negative breathalyzer test
11. Subject is not taking any medications or St. John's wort and agrees to avoid grapefruit juice and alcohol until study completion on Day 28
12. Subject agrees to not take any vitamins or supplements 48 hours prior to dosing
13. Is available for follow-up for the duration of the study

Exclusion Criteria:

1. Received treatment with another investigational drug within 28 days of initial dosing
2. Has a current or history of drug and /or alcohol abuse
3. Is pregnant or breastfeeding woman
4. Has hypersensitivity or allergy to midazolam
5. Has hypersensitivity or allergy to benzodiazepines
6. Has a history of cardiovascular, pulmonary, neurological, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, or psychiatric disease or any other reason, in the opinion of the investigator, that the patient should not participate
7. Tests positive for HIV-1, HIV-2, HbsAg, hepatitis C antibody, or syphilis
8. Has had a blood donation in the 8 weeks prior to the study period start date

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2021-09-17 (Actual)

PRIMARY OUTCOMES:
number of participants with local injection site changes | 28 days
number of participants with systemic changes in physical exam | 28 days
number of participants with vital signs changes resulting in a serious adverse event | 28 days
number of participants with ECG changes resulting in a serious adverse event | 28 days
number of participants with laboratory changes resulting in a serious adverse event | 28 days
time to reach Cmax (Tmax) will be obtained directly from the plasma concentration-time profile data for each patient following IM injection | 28 days
The elimination rate constant (ke) will be estimated | 28 days
The AUC from time 0 to the time of the last measurable concentration (AUC0-last) and the AUC from time zero to infinite time (AUC0-∞) | 28 days

SECONDARY OUTCOMES:
Relative bioavailability will be obtained by analysis of Cmax | 28 days
Relative bioavailability will be obtained by analysis of AUC0-last | 28 days
Relative bioavailability will be obtained by analysis of AUC0-∞ | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Wake Research, Raleigh, North Carolina, United States